CLINICAL TRIAL: NCT02599766
Title: Short-term Effects of Animal-assisted Therapy on the Rehabilitation Process of Brain-injured Patients at REHAB Basel
Brief Title: Effects of Animal-assisted Therapy on Brain-injured Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Institute for Interdisciplinary Research on the Human-Pet Relationship (Other)
Responsible Party: Principal Investigator, Karin Hediger, Dr. phil., Swiss Tropical & Public Health Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ref.Nr.EK:296/13
Record Dates: First submitted 2015-10-29; First posted 2015-11-09 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-04

CONDITIONS: Impaired Social Functioning
Keywords: animal assisted intervention, brain injury, rehabilitation
MeSH Terms: conditions — Brain Injuries | interventions — Animal Assisted Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- animal assisted therapy (Experimental): "Standard therapy" that is done in the presence and with integrating an animal.
  Interventions: Other: animal assisted therapy
- standard therapy (Active Comparator): "Standard therapy" without the presence of an animal.
  Interventions: Other: standard therapy

INTERVENTIONS:
Other: animal assisted therapy — physiotherapy, speech therapy and occupational therapy in the presence of an animal
  Arms: animal assisted therapy
Other: standard therapy — standard physiotherapy, standard speech therapy and standard occupational therapy
  Arms: standard therapy

SUMMARY:
The purpose is to investigate whether animal-assisted therapy has positive biopsychosocial effects on patients with brain injuries. This study investigates the short-term biopsychosocial effects that occur when animals are present during therapy sessions in comparison to therapy sessions without animals, observing a group of 25 patients over 24 therapy sessions. While half of the sessions are held in presence of an animal and half without, they are as comparable as possible with respect to content and setting. In this study, patients who are in a slightly advanced rehabilitation process, assessed via their function profile, are investigated.

DETAILED DESCRIPTION:
This study is designed as a controlled cross-over, within-subject trial with repeated measurement. The experimental condition is the standardised therapy session using therapy animals (AAT), while the control condition is the comparable "standard" therapy session without the presence of an animal.

Over a period of six weeks, patients have four standardised therapy sessions per week, that alternate in a way that two sessions in two consecutive weeks are similar except for one is with the presence of animals and one without. In this way, data is collected over 24 therapy sessions (12 experimental, 12 control) for each patient.

Each therapy session lasts 30 minutes with an additional 5 minutes before and 10 minutes after the session for filling in the questionnaires.

The study takes place at REHAB Basel. Animal-assisted therapies will be held at the "Therapie-Tiergarten" at REHAB Basel in the presence of one or more animals that will be selected by the therapist and the patient together and with which the patient has a relationship.

Patients who are willing to join the study will be selected and allocated randomly to start with either the experimental or the control condition.

Participation in the study will be cancelled if a patient wishes to do so or if they choose to withdraw from the animal-assisted therapy program. Other criteria for withdrawal are if the patient is harmed by an animal or if the animals are abused by the patient.

ELIGIBILITY:
Inclusion Criteria:

* patient at REHAB Basel
* brain-injury
* willing to participate in animal-assisted therapies
* physical and psychological resilience and ability to go/be transported outside to the "Therapie-Tiergarten"
* ability to get in contact with the animal autonomously

Exclusion Criteria:

* medical contraindications:allergies, phobias, etc.
* no willingness to participate in animal-assisted therapies
* patient might present a danger to the animals (aggressive behaviour)
* patient's medication changes radically during the time of data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margret Hund-Georgiadis, PD Dr., Principal Investigator — Rehab Basel
Locations (1):
- REHAB Basel, Basel, Switzerland

REFERENCES:
- [Derived] Gocheva V, Hund-Georgiadis M, Hediger K. Effects of animal-assisted therapy on concentration and attention span in patients with acquired brain injury: A randomized controlled trial. Neuropsychology. 2018 Jan;32(1):54-64. doi: 10.1037/neu0000398. Epub 2017 Oct 16. PMID 29035068

RESULTS

PARTICIPANT FLOW:
Groups:
- AAT and Control Intervention: Animal assisted therapy (AAT): physiotherapy, speech therapy and occupational therapy in the presence of an animal. "Standard therapy" that is done in the presence and with integrating an animal.
  Duration of AAT: 6 weeks (12 AAT sessions) Frequency of administration: 2 sessions/week
  Control intervention: standard therapy (treatment as usual): physiotherapy, speech therapy and occupational therapy without an animal Duration of control therapy: 6 weeks (12 sessions) Frequency of administration: 2 sessions/week
Period: Overall Study
Arm/Group | AAT and Control Intervention
Started | 22
Completed | 19
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- AAT and Control Intervention: Animal assisted therapy (AAT): physiotherapy, speech therapy and occupational therapy in the presence of an animal
  Control intervention: standard physiotherapy, speech therapy and occupational therapy
Arm/Group | AAT and Control Intervention
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.84 (14.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 19
FIM (Functional Independence Measure) [Mean (Standard Deviation); unit: units on a scale] — The FIM includes 18 items, each with a maximum score of 7 and a minimum score of 1. Possible scores range from 18 to 126. Each level of scoring is defined with higher scores refering to better outcomes.
  units on a scale | 68.67 (26.08)

OUTCOME MEASURES:

1. Primary Outcome: Social Functioning: Total Social Behavior
Description: Interaction and communication behavior is assessed via video coding in Noldus Observer. Percentage of all social behaviors are collected and aggregated to one measure, the total social behavior.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of shown behavior
Arm/Group | Animal Assisted Therapy | Standard Therapy
Number analyzed (Participants) | 19 | 19
percentage of shown behavior | 29.22 (15.66) | 8.68 (8.85)

2. Secondary Outcome: Social Functioning: Verbal Communication
Description: Interaction and communication behavior is assessed via video coding in Noldus Observer. Percentages of the defined verbal behaviors is collected and aggregated to one measure.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of verbal communication
Groups:
- Animal Assisted Therapy: Animal assisted therapy (AAT): physiotherapy, speech therapy and occupational therapy in the presence of an animal. "Standard therapy" that is done in the presence and with integrating an animal.
  Duration of AAT: 6 weeks (12 AAT sessions) Frequency of administration: 2 sessions/week
- Control Intervention: Control intervention: standard therapy (treatment as usual): physiotherapy, speech therapy and occupational therapy without an animal Duration of control therapy: 6 weeks (12 sessions) Frequency of administration: 2 sessions/week
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
percentage of verbal communication | 25.4 (19.44) | 19.04 (20.24)

3. Secondary Outcome: Social Functioning: Nonverbal Communication
Description: Interaction and communication behavior is assessed via video coding in Noldus Observer. Percentage of the defined nonverbal behaviors is collected and aggregated to one measure.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of nonverbal communication
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
percentage of nonverbal communication | 31.94 (17.54) | 5.26 (7.09)

4. Secondary Outcome: Social Functioning: Physical Contact
Description: Interaction and communication behavior is assessed via video coding in Noldus Observer. Percentage of the defined physical contact is collected and aggregated to one measure.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of physical contact
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
percentage of physical contact | 18.32 (18.50) | 1.53 (9.70)

5. Secondary Outcome: Social Functioning: Attention
Description: Interaction and communication behavior is assessed via video coding in Noldus Observer. Percentage of the defined attention behavior is collected and aggregated to one measure.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: percentage of attention
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
percentage of attention | 89.01 (2.01) | 90.65 (2.00)

6. Secondary Outcome: Positive Emotional Display
Description: Emotional display is assessed via video coding in Noldus Observer. Percentage of the defined behavior during the therapy sessions is collected and aggregated to one measure of positive emotion.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of positive emotion
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
percentage of positive emotion | 6.95 (7.47) | 3.75 (4.57)

7. Secondary Outcome: Negative Emotional Display
Description: Emotional display is assessed via video coding in Noldus Observer. Percentage of the defined behavior during the therapy sessions is collected and aggregated to one measure of negative emotion.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of negative emotion
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
percentage of negative emotion | 0.31 (1.34) | 0.59 (2.05)

8. Secondary Outcome: Neutral Emotional Display
Description: Emotional display is assessed via video coding in Noldus Observer. Percentage of the defined behavior during the therapy sessions is collected and aggregated to one measure of neutral emotion.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of neutral emotion
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
percentage of neutral emotion | 92.73 (7.64) | 94.20 (6.60)

9. Secondary Outcome: Mood 1: Motivation
Description: Assessed via visual analogue scale as self-rating Scale ranging from 0 (not motivated) to 160 (highly motivated)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
units on a scale | 138.80 (27.13) | 132.22 (28.21)

10. Secondary Outcome: Mood 2: Bipolar Mood Dimension (Good-bad)
Description: Assessed via the Mehrdimensionaler Befindlichkeitsfragebogen (MDBF) We analysed the bipolar mood dimension (good-bad) ranging from 4 (not at all good mood) to 20 (very good mood).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
units on a scale | 16.93 (4.20) | 16.12 (4.29)

11. Secondary Outcome: Mood 3: Satisfaction Self-assessment
Description: Assessed via visual analogue scale as rating by the therapist Satisfaction during the therapy sessions was assessed by the patient themselves using a VAS ranging from 0 (unsatisfied) to 160 (satisfied).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
units on a scale | 129.81 (23.80) | 124.54 (37.81)

12. Secondary Outcome: Mood 4: Satisfaction Therapist Rating
Description: Satisfaction during the therapy sessions was assessed by the therapist using a VAS ranging from 0 (unsatisfied) to 160 (satisfied).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
units on a scale | 137.31 (23.80) | 128.14 (27.75)

13. Secondary Outcome: Heart Rate
Description: Assessed via EKG (Polar) during the sessions and measured in beat/min.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
beats per minute | 85.23 (13.03) | 83.41 (14.86)

14. Secondary Outcome: Motor Activity
Description: Assessed via actimeter at the patients wrist during sessions, measuring acceleration of the hand. It records data in 15-s epochs for maximum sensitivity. Data were calculated to yield average activity Counts per minute.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: counts per minute
Arm/Group | Animal Assisted Therapy | Control Intervention
Number analyzed (Participants) | 19 | 19
counts per minute | 90.93 (55.45) | 75.88 (60.67)

ADVERSE EVENTS:
Time Frame: Through study completion, 6 weeks
Arm/Group | Animal Assisted Therapy | Standard Therapy
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No